CLINICAL TRIAL: NCT00634608
Title: Integrating Targeted MedlinePlus Health Prescriptions Into Clinic Practice Workflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HHSN276200700263P
Record Dates: First submitted 2008-02-22; First posted 2008-03-13 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Allergic Rhinitis; Asthma; Back Pain; Benign Prostatic Hypertrophy; Bursitis; Depression; Anxiety; Diabetes Mellitus; Esophageal Reflux; HIV Infections; Hyperlipidemia; Hypertension; Insomnia; Irritable Bowel Syndrome; Obesity; Osteoporosis (Senile); Shoulder Pain; Sinusitis; Symptomatic Menopause; Urinary Incontinence; Urinary Tract Infection; Vaginitis
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Back Pain; Prostatic Hyperplasia; Bursitis; Depression; Anxiety Disorders; Diabetes Mellitus; Gastroesophageal Reflux; HIV Infections; Hyperlipidemias; Hypertension; Sleep Initiation and Maintenance Disorders; Irritable Bowel Syndrome; Obesity; Osteoporosis; Shoulder Pain; Sinusitis; Urinary Incontinence; Urinary Tract Infections; Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Survey (No Intervention): Control group participants are sent a survey within one week of clinic visit
- Health Information Prescription (Experimental): Health Information Prescription is emailed to participants within 24 hours of clinic visit.
  Interventions: Other: Health Information Prescription

INTERVENTIONS:
Other: Health Information Prescription — The patient education materials will consist of approximately 21 topics representing some of the most common conditions seen at the Fairview Internal Medicine Clinic. Twenty-one e-mails, one per topic, will be created by Fairview physicians to be distributed to selected clinic patients. There will be a standard e-mail for each condition with a specific link to MedlinePlus. To create the targeted health information topic email, the physician will review the information available at MedlinePlus. The physician will then select several links of appropriate information and, using the template, will write a short annotation on each link.
  Arms: Health Information Prescription

SUMMARY:
The specific aim of this proposed project is to implement a standard process for integrating MedlinePlus health information prescriptions into the clinic workflow.

Hypothesis 1: Individuals in the intervention group who receive tailored email health information with provider selected MedlinePlus links and added commentary for patient specific conditions will be more likely to seek information / use MedlinePlus compared with individuals in the control group.

Hypothesis 2: Individuals in the intervention group who receive tailored email health information with provider selected MedlinePlus links and added commentary for patient specific conditions will be more satisfied with the information received compared with individuals in the control group.

DETAILED DESCRIPTION:
Providing patient education in an outpatient practice can be challenging in part due to the variety of patient medical conditions and the quantity of materials needed. Increasingly, electronic resources such as those found on the internet have the potential to provide easily accessible needed information. However, clinicians do not have the time to assemble a list of websites for their patients and even if they did, the quality of information varies greatly and would require close screening. MedlinePlus is a free National Library of Medicine sponsored website that features health information on hundreds of conditions with all information carefully screened for quality standards by expert librarians. We will conduct a pilot study to seamlessly integrate provider-customized MedlinePlus health education prescriptions for specific conditions into the normal clinic workflow to motivate patients to access and expand their use of MedlinePlus to benefit their health. As HIV prevention/education is very important, we will include the HIV clinic as well as a general internal medicine clinic.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study population, patients must also be seen by their physician for one of the 21 target health conditions (Allergic Rhinitis, Asthma, Back Pain, Benign Prostatic Hypertrophy, Bursitis, Depression/Anxiety, Diabetes Mellitus, Esophageal Reflux, HIV, Hyperlipidemia, Hypertension, Insomnia, Irritable Bowel Syndrome, Obesity, Osteoporosis (senile), Shoulder Pain, Sinusitis, Symptomatic Menopause, Urinary Incontinence, Urinary Tract Infection, Vaginitis) and be willing to provide an email address.
* Patients will be included only once.
* All patients in the intervention and the control group will receive the survey.
* All physicians and staff at the Fairview Clinic and HIV Clinic will be invited to complete the physician or staff survey.

Exclusion Criteria:

* No email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
health information experiences of the patient | approximately one week following clinic appointment

SECONDARY OUTCOMES:
clinician feedback on the health information prescription process | midpoint and conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hodge, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Department of Internal Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coberly E, Boren SA, Davis JW, McConnell AL, Chitima-Matsiga R, Ge B, Logan RA, Steinmann WC, Hodge RH. Linking clinic patients to Internet-based, condition-specific information prescriptions. J Med Libr Assoc. 2010 Apr;98(2):160-4. doi: 10.3163/1536-5050.98.2.009. No abstract available. PMID 20428282